CLINICAL TRIAL: NCT00000326
Title: Buprenorphine/Naloxone Treatment for Opioid Dependence-Experiment 1(1)
Brief Title: Buprenorphine/Naloxone Treatment for Opioid Dependence-Experiment 1 - 1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-11160-1; 1R01DA011160 (NIH); R01-11160-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: Heroin Dependence
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders

INTERVENTIONS:
Drug: Heroin Dependence

SUMMARY:
The purpose of this study is to assess the clinical efficacy of the buprenorphine/naloxone combination tablet for alternate-day dosing and determine whether multiples of the daily dose are necessary to maintain an effective alternate day dosing regimen.

DETAILED DESCRIPTION:
Alternate-day dosing with the 8mg buprenorphine-naloxone tablet is as safe and effective as daily dosing. Outcomes are improved when the total weekly dose provided during alternate-day dosing is equal to that given during daily dosing.

ELIGIBILITY:
Inclusion Criteria:

Individuals must be currently opioid dependent and meet FDA criteria for narcotic maintenance treatment. Co-morbid substance abuse or dependence disorders may also be present. Individuals must be healthy despite drug dependency.

Exclusion Criteria:

Individuals with evidence of an active Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Axis I psychiatric disorder (e.g. psychosis, manic-depressive illness, organic psychiatric disorders), significant medical illness (e.g. liver or cardiovascular disease) or pregnant female subjects are excluded from study participation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 1997-04; Primary Completion 1997-08 (Actual); Study Completion 1997-08 (Actual)

PRIMARY OUTCOMES:
Drug use
Retention
Subjective dose estimate
Observed withdrawal rating
Opioid agonist rating
Opioid antagonist rating
Pupil diameter
Compliance
Analog rating scale for drug effects
Drug effect characteristics
Dose order estimate-nurse
Dose order estimate-client

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Amass, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Background] (presented at ACNP 1997. Kamien, J.B., Mikulich, S.K., and Amass, L., Efficacy of the buprenorphine/naloxone tablet for daily vs. alternate-day opioid dependence treatment. Presented to the 1998 Meeting of the College on Problems of Drug Dependence.. Presented at ACNP 1997 and CPDD 1998.